CLINICAL TRIAL: NCT02524002
Title: Clear Liquids vs Enhanced Clear Liquids; Effect on Labor Performance
Brief Title: Enhanced vs. Routine Clear Liquid Intake in Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 22375
Record Dates: First submitted 2014-08-15; First posted 2015-08-14 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Abnormal Labor; Failed Induction of Labor; Ketosis
Keywords: Abnormal Labor; Prolonged Induction; Ketosis; Diet
MeSH Terms: conditions — Dystocia; Ketosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Clear Diet (Placebo Comparator): This intervention consists of soup broth, variety of juices (apple, cranberry, grape), ginger ale, water, and ice.
  Interventions: Dietary Supplement: Usual clear diet
- Accel Gel (Experimental): This intervention is an enhanced clear liquid gel is Accel Gel, produced by PacificHealth Labs of Matawan, NJ. This gel has 4:1 carb to protein ratio formula, and ingredients that are not contraindicated in pregnancy (only the flavors with minimal caffeine are used).
  http://www.pacifichealthlabs.com/accel-gel-all-natural-rapid-energy-gel-product.html
  Interventions: Dietary Supplement: Accel Gel

INTERVENTIONS:
Dietary Supplement: Accel Gel — Accel Gel by PacificHealth Labs in Matawan, NJ.
  Arms: Accel Gel
Dietary Supplement: Usual clear diet — Usual clear liquids
  Arms: Usual Clear Diet

SUMMARY:
The goal of the study is to see if the addition of a carbohydrate- and protein-enhanced gel during labor speeds labor and reduces the rate of cesarean delivery.

DETAILED DESCRIPTION:
Patients will be randomized to placebo or experimental arm of study. In the placebo arm, patients will receive standard clear liquid diet, which includes ginger ale, variety of fruit juices, and plain soup broth. The experimental arm will receive the standard clear liquid diet, and in addition will receive Accel Gel every 3 hours while in labor.

ELIGIBILITY:
Inclusion criteria:

* Nulliparity (first baby)
* Admission with the intent to deliver vaginally
* Gestational age >36 weeks
* Age ≥ 18

Exclusion criteria:

* Planned cesarean delivery
* Renal Disease
* Preeclampsia
* Diabetes (Pre-gestational or Gestational)
* Allergy to any component of sports drink
* NPO diet by physician

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2014-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Time from admission to delivery | Participants will be followed during labor until delivery, an expected range of 1-48 hours
  Up to 3 days from time of admission

SECONDARY OUTCOMES:
Duration of second stage of labor | Participants will be followed during labor until delivery, an expected range of 1-48 hours
  Time of complete cervical dilation to delivery of infant
delivery in <24 hours | Participants will be followed during labor until delivery, an expected range of 1-48 hours
cesarean delivery | Participants will be followed during labor until delivery, an expected range of 1-48 hours
rate of composite adverse GI outcome (vomiting or diarrhea) | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  Any vomiting or diarrhea
patient satisfaction with diet | Participants will be followed during labor until delivery, an expected range of 1-48 hours
Urine Ketones | Participants will be followed during labor until full dilation, an expected range of 1-48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Laura Goetzl, M.D., Principal Investigator — Temple University Hospital
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes